CLINICAL TRIAL: NCT04595942
Title: Comparison of Outcomes With Midodrine and Fludrocortisone for Objective Recurrence in Treating Syncope (COMFORTS Trial)
Brief Title: Midodrine and Fludrocortisone for Vasovagal Syncope
Acronym: COMFORTS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran Heart Center (Other)
Collaborators: Mahidol University (Other); Rajaie Cardiovascular Medical and Research Center (Other); Tehran Arrhythmia Center (Unknown); Imam Khomeini Hospital (Other); AJA University of Medical Sciences (Other); Urmia University of Medical Sciences (Other); Isfahan University of Medical Sciences (Other); Shahid Beheshti University of Medical Sciences (Other); Ahvaz Jundishapur University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Masih Tajdini, MD, Assistant Professor of Cardiology, Tehran Heart Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 99-2-408-49493
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Syncope, Vasovagal
Keywords: Syncope, Vasovagal; Syncope; Midodrine; Fludrocortisone; Randomized Controlled Trial
MeSH Terms: conditions — Syncope, Vasovagal; Syncope | interventions — Midodrine; fludrocortisone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Midodrine (Active Comparator): 10 mg midodrine three times a day
  Interventions: Drug: Midodrine Hydrochloride Tablets; Behavioral: Lifestyle modification
- Fludrocortisone (Active Comparator): 0.1 mg fludrocortisone two times a day
  Interventions: Drug: Fludrocortisone Acetate Tablets; Behavioral: Lifestyle modification
- Lifestyle modification (Other): Education, salt and water intake, counter-pressure maneuvers
  Interventions: Behavioral: Lifestyle modification

INTERVENTIONS:
Drug: Midodrine Hydrochloride Tablets — Patients will be started on 5 mg Midodrine three times a day and after one week the dosage will be up-titrated to 10 mg three times a day and continued for 12 months. They will receive the medication at four-hour intervals upon rising in the morning (the last dose should not be taken later than 6 PM). In case of intolerance, the dosage will be reduced to 2.5 mg three times a day. Patients will also receive recommendations for lifestyle modifications including drinking 2 to 3 liters of fluid per day, daily consumption of 10 grams of salt, and practicing counter-pressure maneuvers (handgrip, arm-tensing, leg crossing and squatting).
  Other Names: Gutron
  Arms: Midodrine
Drug: Fludrocortisone Acetate Tablets — Patients will be started on 0.05 mg of fludrocortisone twice daily and after one week the dosage will be up-titrated to 0.1 mg fludrocortisone twice daily taken for 12 months. Patients will also receive recommendations for lifestyle modifications including drinking 2 to 3 liters of fluid per day, daily consumption of 10 grams of salt, and practicing counter-pressure maneuvers (handgrip, arm-tensing, leg crossing and squatting). In this arm, potassium levels will be checked 7-14 days after dose stabilization.
  Other Names: Florinef
  Arms: Fludrocortisone
Behavioral: Lifestyle modification — Patients will be recommended to drink 2 to 3 liters of fluid per day, consume 10 grams of salt per day, and practice counter-pressure maneuvers (handgrip, arm-tensing, leg crossing and squatting) for 12 months.

SUMMARY:
Syncope is a common condition which can disturb daily functions of the patients and impair their quality of lives. It contributes to 0.8 to 2.4% of the visits of emergency rooms. Noticeably, studies demonstrated that the lifetime prevalence of syncope is as high as 41% with a 13.5% recurrence rate.

The cornerstone of the treatment of vasovagal syncope (VVS), the most common type of syncope, is lifestyle modifications and patient education to avoid potential triggers of syncope. These recommendations alleviate vasovagal spells in many patients; however, some patients experience life-disturbing vasovagal attacks despite compliance with these modifications. This fact underscores the importance of efficient pharmacological interventions as well.

Currently, there is an ongoing controversy about the efficacy of midodrine and fludrocortisone as adjunct pharmacological interventions for the prevention of VVS. In the COMFORTS trial, we are going to evaluate the efficacy of midodrine, fludrocortisone, and lifestyle modifications for prevention of vasovagal attacks in patients with VVS.

DETAILED DESCRIPTION:
Background: The cornerstone of the treatment of vasovagal syncope (VVS) is lifestyle modifications; however, some patients incur life-disturbing attacks despite compliance with these treatments which underscores the importance of pharmacological interventions.

Methods: In the COMFORTS trial, a multi-center randomized controlled trial, 1375 patients with VVS will be randomized into three parallel arms with a 2:2:1 ratio to receive midodrine, fludrocortisone, or just lifestyle modifications. All patients will receive recommendations for lifestyle modifications. In the pharmacological intervention arms, patients will receive 5 mg of midodrine three times a day or 0.1 mg of fludrocortisone twice daily. In case of intolerance, the dosage will be cut by half. If the patient does not tolerate even the reduced dosage, the medication will be discontinued and the patient will be advised to use compression garments, practice tilt training exercises, or switch to the other medication. The patients will be followed on 3, 6, and 12 months after dose stabilization. Primary efficacy outcomes of the study is the time to the first syncopal episode. The secondary efficacy outcome are the recurrence rate of syncope, number of syncopal episodes and the quality of life of the patients which will be assessed by the 36-Item Short Form Survey questionnaire at the enrollment and 12 months after dose stabilization.

ELIGIBILITY:
Inclusion Criteria:

* Vasovagal syncope as the cause of transient loss of consciousness (Clinical diagnosis AND Calgary Syncope Symptom Score ≥ -2; Head-up tilt test is not mandatory for diagnosis)
* ≥2 episodes of syncope during the last year
* Medication-naïve or have at least a 2-week washout period prior to randomization
* The capability of giving informed consent
* Signed written informed consent

Exclusion Criteria:

* Other causes of transient loss of consciousness including orthostatic hypotension, postural tachycardia, carotid sinus hypersensitivity, or seizure
* Cardiac rhythm disorders including ventricular tachycardia, long QT syndrome, Brugada syndrome, arrhythmogenic right ventricular cardiomyopathy, complete heart block, and any conduction abnormality on electrocardiogram
* Severe valvular heart disease
* Hypertrophic cardiomyopathy
* Cardiac systolic dysfunction (ejection fraction≤40%)
* Obstructive coronary artery disease
* Hypertension
* Diabetes mellitus
* Cirrhosis
* Renal failure stage≥3
* Known intolerance or hypersensitivity to midodrine or fludrocortisone
* Urinary retention
* Pheochromocytoma
* Thyrotoxicosis
* Glaucoma
* Previous use of midodrine or fludrocortisone for treatment of VVS or another condition
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1375 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Time to first episode of syncope | The follow-up continues for 12 months after randomization
  Time from randomization to occurrence of the first episode of vasovagal syncope during the follow-up.

SECONDARY OUTCOMES:
Recurrence rate of vasovagal syncope | The follow-up continues for 12 months after randomization
  The proportion of patients who incurred at least one episode of vasovagal syncope during the follow-up.
Changes in quality of life | Baseline (It will be evaluated at randomization) and 12 months after randomization.
  It is measured by the 36-item short form (SF-36) questionnaire.
Major side effects | The follow-up continues for 12 months after randomization
  The proportion of patients who do not tolerate the initial dosage of medications which leads to either a reduced dosage or discontinuation.
Minor side effects | The follow-up continues for 12 months after randomization
  The proportion of patients who experience minor side effects without dosage changes.

CONTACTS AND LOCATIONS:
Overall Officials: Arash Jalali, PhD, Study Director — Tehran Heart Center, Tehran University of Medical Sciences; Arya Aminorroaya, MD, MPH, Study Director — Tehran Heart Center, Tehran University of Medical Sciences; Hamed Tavolinejad, MD, Study Director — Tehran Heart Center, Tehran University of Medical Sciences; Saeed Sadeghian, MD, Study Chair — Tehran Heart Center, Tehran University of Medical Sciences
Locations (1):
- Tehran Heart Center, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No
The data is not publicly available due to privacy/ethical restrictions. The data can be shared upon reasonable request to the trial committee,

REFERENCES:
- [Background] Aminorroaya A, Tavolinejad H, Sadeghian S, Jalali A, Alaeddini F, Emkanjoo Z, Mollazadeh R, Bozorgi A, Oraii S, Kiarsi M, Shahabi J, Akbarzadeh MA, Rahimi B, Joharimoghadam A, Mohsenizade A, Mohammadi R, Oraii A, Ariannejad H, Apakuppakul S, Ngarmukos T, Tajdini M. Comparison of Outcomes with Midodrine and Fludrocortisone for Objective Recurrence in Treating Syncope (COMFORTS trial): Rationale and design for a multi-center randomized controlled trial. Am Heart J. 2021 Jul;237:5-12. doi: 10.1016/j.ahj.2021.03.002. Epub 2021 Mar 6. PMID 33689731
- [Background] Sadeghian S, Aminorroaya A, Tajdini M. The Syncope Unit of Tehran Heart Center. Eur Heart J. 2021 Jan 7;42(2):148-150. doi: 10.1093/eurheartj/ehaa532. No abstract available. PMID 33346809